CLINICAL TRIAL: NCT07010575
Title: Decentralized Study to Assess Patient Treatment Preference Comparing Their Current Standard-of-care Wilson's Disease (WD) Treatment to a New Trientine (TETA) 4HCl Formulation.
Brief Title: Patient Preference Study: Standard of Care Versus Once-daily Trientine Tetrahydrochloride
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orphalan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORPH-131-015
Record Dates: First submitted 2025-05-12; First posted 2025-06-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Once Daily Administration of new TETA 4HCl followed by return to standard of care (Experimental): The new formulation of TETA 4HCl will be administered once a day for 28 days. Each film-coated tablet contains 300 mg of trientine base.
  Once completed patients will return to their standard of care Wilson's Disease treatment and be followed for a further 28 days.
  Interventions: Drug: New TETA 4HCl Formulation; Drug: Standard of Care

INTERVENTIONS:
Drug: New TETA 4HCl Formulation — Individual patient doses will depend on the Standard of Care (SOC) therapy at study entry and guided by recommended dosing switch schedule outlined in the study protocol. The dose may subsequently be titrated based on clinical response per the investigator's judgement.
Drug: Standard of Care — Patients will be returned to their approved Wilson's Disease SOC therapy (dose and frequency) at study entry as prescribed by their treating Wilson's Disease physician.

SUMMARY:
Decentralized study to assess patient reported treatment satisfaction comparing their current standard-of-care Wilson's Disease (WD) treatment with a new once-daily Trientine (TETA) 4HCl formulation.

DETAILED DESCRIPTION:
This is a single arm study where patients on Standard of Care maintenance therapy with a prescribed approved Wilson's Disease therapy administered at least twice daily will be screened for eligibility by the clinical research site either following referral from a participant identification centre (PIC) or following advertisements. An initial screening Patient Reported Outcome (PRO) assessment including the Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) and Morisky Medication Adherence Scale-8 (MMAS-8) will also be collected.

Patients who meet all the study entry criteria will be switched to a new TETA 4HCl formulation for 28 days and will be monitored using Patient Reported Outcomes and specific posology questions held within a patient questionnaire pack and blood investigations. During this treatment phase (between Day 14 and Day 28 of dosing), each participant will be interviewed to collect qualitative data on disease and therapy. Patients will then be returned to their Standard of Care treatment and followed for a further 28 days continuing to be assessed using Patient Reported Outcomes and repeat blood investigations. The safety period will be finalised with an End of Study Assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent for participation in the study.
2. Proficient and fluent in English language speaker, writer and reader.
3. Patients of any gender, aged 18 years or older as of signing the Informed Consent Form (ICF).
4. Patients on current SOC WD maintenance treatment prescribed twice daily (or more frequently) and dose has been unchanged for at least 3-months.
5. Women of childbearing potential and sexually active males must agree to adhere to a contraceptive method.

Exclusion Criteria:

1. Major systemic disease or other illness that would, in the opinion of the investigator, compromise patient safety or interfere with the collection or interpretation of the study results.
2. Patients with severe anaemia (e.g., Haemoglobin <10 g/dL).
3. Female participants who are pregnant (including a positive pregnancy test at Screening and on Day-1) or breastfeeding.
4. Any contraindications as described in the current Investigator Brochure for TETA 4HCl.
5. Subject receiving total daily dose of chelator as SOC greater or equal to 1200mg (trientine base or d-penicillamine).
6. In the opinion of the investigator, the patient is likely to be a non-attender or uncooperative for routine clinical visits during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Assess and compare patient preference, convenience and satisfaction between current standard of care treatments for Wilson's Disease and the new TETA 4HCl formulation using patient reported outcome questionnaires. | From the screening assessment (-28 days to Day 1) to end of study at Week 8
  Mean Treatment Satisfaction Questionnaire for Medication (TSQM-9) score over time including change from baseline by domain
Assess and compare patient preference, convenience and satisfaction between current standard of care treatments for Wilson's Disease and the new TETA 4HCl formulation using patient reported outcome questionnaires. | From the screening assessment (-28 days to Day 1) to end of study at Week 8
  Incidence of categorical posology questions over time

SECONDARY OUTCOMES:
Assess treatment adherence and tolerability of a new TETA 4HCl formulation. | From the screening assessment (-28 days to Day 1) to end of study at Week 8
  Mean Morisky Medication Adherence Scale-8 (MMAS-8) score over time including change from baseline
Assess treatment adherence and tolerability of a new TETA 4HCl formulation. | From the screening assessment (-28 days to Day 1) to end of study at Week 8
  Incidence of categorical laboratory safety data and adverse events (AE) assessments during the study.
Assess treatment adherence and tolerability of a new TETA 4HCl formulation. | From the screening assessment (-28 days to Day 1) to end of study at Week 8
  Mean of continuous laboratory safety data during the study

OTHER OUTCOMES:
Assess markers of copper balance with a new TETA 4HCl formulation. | From the screening assessment (-28 days to Day 1) to end of study at Week 8
  Mean Serum NCC values as assessed by speciation assay (NCC-Sp);
Qualitative data analysis following a semi-structured patient interview designed to develop a WD-specific PRO measure. | From Day 14 to Day 28
  Cognitive validation of a novel Wilson's disease-specific patient reported outcome measure under development using qualitative patient interview data on disease and therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Davidsson, Principal Investigator — VCTC
Locations (1):
- VCTC, Hartshorne, Derbyshire, United Kingdom